CLINICAL TRIAL: NCT07062692
Title: Effectiveness of Dry Needling Versus Manual Trigger Point Release on Active Rhomboid Trigger Points
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01017 Khaist Yousafzai
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Rhomboid Trigger Points
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needling trigger release therapy (Experimental): This group will undergo dry needling trigger release therapy. Total of 2 sessions (one per week) followed by home based exercises plan. Treatment protocol of both groups will include Therapeutic ultrasound, Cold pack application and Home based exercise plan.
  Interventions: Other: dry needling trigger release therapy
- MANUAL TRIGGER POINT RELEASE (Experimental): Manual trigger release will be given to the other group. Total of 2 sessions (one per week) followed by same home based exercises plan will be given to the both groups. Treatment protocol of both groups will include Therapeutic ultrasound, Cold pack application and Home based exercise plan.
  Interventions: Other: MANUAL TRIGGER POINT RELEASE

INTERVENTIONS:
Other: dry needling trigger release therapy — The dry needling intervention involved inserting sterile filiform needles directly into active rhomboid trigger points for 1-2 sessions (1 session/week) to elicit local twitch responses and relieve tension.
  Arms: dry needling trigger release therapy
Other: MANUAL TRIGGER POINT RELEASE — The manual trigger point release intervention involved applying sustained pressure to active rhomboid trigger points followed by passive stretching to release muscle tension and improve mobility.
  Arms: MANUAL TRIGGER POINT RELEASE

SUMMARY:
This study compares dry needling and manual trigger point release for treating active rhomboid trigger points in 48 patients, assessing pain, ROM, and function. It addresses a gap in evidence for optimal pain management in upper back myofascial pain. Findings will guide clinical practice for more effective, evidence-based interventions.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) investigates the effectiveness of dry needling versus manual trigger point release in treating active rhomboid trigger points. The study aims to compare the effect of two interventions on pain, range of motion (ROM), and functional outcomes in patients with rhomboid muscle pain.

Participants: 48 individuals (aged 20-60) with clinically confirmed active rhomboid trigger points.

Interventions:

Group 1: Dry needling therapy.

Group 2: Manual trigger point release. Both groups receive adjunct therapies (ultrasound, cold packs, and home exercises).

Outcome Measures: Pain (Numeric Pain Rating Scale), ROM (goniometer), and function (DASH Questionnaire).

Duration: 2-week intervention with follow-ups at 1 and 2 weeks.

Significance: The study addresses a gap in evidence for rhomboid trigger point treatments, guiding clinical decisions for pain management. Results may optimize therapeutic approaches for upper back pain.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a clinically confirmed active trigger point in the rhomboid muscle based on established criteria (e.g., palpable tight band, local tenderness, referred pain pattern).
* Pain Level: Moderate to severe pain intensity (e.g., 4 or higher on a Visual Analog Scale or Numeric Pain Rating Scale).
* Duration of Symptoms: pain for at least 4 weeks.

Exclusion Criteria:

* Patient with conditions that may contribute to neck and subscapular pain other than rhomboid:
* fibromyalgia
* Rheumatic and inflammatory disease
* Recent Surgery
* Diabatic
* Cervical radiculopathy and nerve entrapment
* Pregnancy
* Malignancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-23 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 2 Weeks
  A subjective pain assessment tool where patients rate their pain intensity on a scale from 0 (no pain) to 10 (worst imaginable pain).
Goniometer | 2 Weeks
  The goniometer is a handheld device with a protractor and movable arms used to precisely measure joint range of motion in degrees.
DASH Questionnaire | 2 Weeks
  The DASH Questionnaire is a 30-item self-report tool assessing upper extremity function and symptoms in daily activities, scored from 0 (no disability) to 100 (severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Amna Anum, ms, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Malakand, Chakdara, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No